CLINICAL TRIAL: NCT06436404
Title: Effect of Two Different Positions on Pain, Stress, Comfort and Physiological Parameters of the Premature Infants: Randomized Controlled Trial
Brief Title: Hammock Position and Kangaroo Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: He2
Record Dates: First submitted 2024-05-08; First posted 2024-05-31 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-12

CONDITIONS: Infant Development; Premature
Keywords: Premature; Pain; Stress; Comfort
MeSH Terms: conditions — Premature Birth; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled, single-blind parallel design experimental study.In the study, premature infants will be divided into three groups by randomization.
  Each group will be referred to as A, B or C for convenience.
  The type of intervention will be determined by drawing lots for A, B and C.
  For example, A= Hammock Position, B= Kangaroo Care c=Control Group.
  When applying the hammock position to a group; The other group will receive kangaroo care, while the other group will receive standard care.
  For randomization, blocks of 3 created for 42 infants and this process done by an independent statistician.
Who Masked: Participant
Masking Description: Single blinding (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hammock position group (Experimental): A hammock inside the incubator, developed by researchers to prevent heat loss and support posture, will be used.
  Interventions: Other: Hammock intervention
- Kangaroo care group (Experimental): Kangaroo care will be applied to these preterm infants.
  Interventions: Other: Kangaroo care intervention
- Contol group (No Intervention): The group will not receive any other intervention.

INTERVENTIONS:
Other: Hammock intervention — It is a hammock made of 100% cotton fabric that prevents heat loss and has an internal apparatus to support the position, which can be adapted to the incubator by the researchers.
  Arms: Hammock position group
Other: Kangaroo care intervention — In the clinic, the baby will receive kangaroo care with his mother in a quiet room with reduced lighting.
  Arms: Kangaroo care group

SUMMARY:
This study was planned to evaluate the effectiveness of two positions that may have an effect on pain, stress, comfort and physiological parameters in premature infants.

DETAILED DESCRIPTION:
Providing adequate therapeutic positioning in preterms can minimize postural abnormalities and asymmetries associated with prematurity and NICU stay, as well as support the development of spontaneous and functional motor abilities of infants. Studies show that positioning directly affects cardiovascular, respiratory and sleep-wake states. When the literature is examined; Although the vital signs, pain levels and comfort levels of babies in the NICU have been examined in many applications, the number of studies comparing the hammock position and Kangaroo care in preterms is very limited. Therefore, this study will try to determine the effect of hammock position and kangaroo care on the pain, stress, comfort and physiological parameters of the infants. It is thought that the study will provide new data to the literature and lead to many researches.

ELIGIBILITY:
Inclusion Criteria:

* Infants having at least 2 days of inpatient treatment from,
* Infants 32-36+6. being born during the gestational week,
* Infants not receiving a medical diagnosis other than prematurity (serious respiratory, cardiological, endocrine and metabolic problems, hearing problems, hypoglycemia and sepsis),
* Apgar score above 6 at the 5th minute Infants will included.

Exclusion Criteria:

* Infants having at least 2 days of inpatient treatment from,
* Infants 32-36+6. being born during the gestational week,
* Infants not receiving a medical diagnosis other than prematurity (serious respiratory, cardiological, endocrine and metabolic problems, hearing problems, hypoglycemia and sepsis),
* Apgar score above 6 at the 5th minute Infants will included.

Ages: 32 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Determining the descriptive characteristics of babies | 1 hour
  1- Infant Introductory Form: The form includes introductory information about the baby (Postnatal day, gestational age, birth weight (g), weight on the day of the intervention, type of birth, gender, postnatal age, physiological weight loss, feeding style, 1st and 5th minute Apgar score, maternal age. It consists of questions containing).
Hammock position and Kangaroo care increase comfort level in preterm infants | 1 hour
  2- The COMFORT-behavior scale (COMFORTneo): It is a Likert-type scale developed to be used in evaluating the sedation and comfort needs, pain and distress of newborns monitored in intensive care. The scale was revised for newborns. High scores indicate that the baby is not comfortable and needs interventions to provide comfort.
Hammock position and Kangaroo care decrease pain and stress level in preterm infants | 1 hour
  3- ALPS-Neo "Newborn Pain and Stress Assessment Scale": The scale was developed in 2014 to evaluate pain and stress in premature and term newborns. Measurement is made through observation. As the score obtained increases, stress and pain increase.

SECONDARY OUTCOMES:
Hammock position and Kangaroo care support physiological stability in premature infants. | 1 hour
  1- Physiological Parameter Tracking Chart The follow-up chart prepared by the researcher is a form in which physiological parameters such as heart rate (min), oxygen saturation (%SpO2), body temperature (°C), respiratory rate (min) are recorded. Measurements will be taken 3 times in total: before, during and after the hammock position and kangaroo care application. A monitor device used in clinical routine will be used to measure physiological parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel KUCUKOGLU, Ph.D., Study Director — Selcuk University; Halil DEGIRMENCIOGLU, Md., Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Niğde Ömer Halisdemir University, Niğde, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Indyk HE, Woollard DC. Enzymatic determination of free carnitine in milk and infant formulas. J AOAC Int. 1995 Jan-Feb;78(1):69-74. PMID 7703730
- [Background] Costa KSF, Fernandes DDS, Paula RAP, Guarda LEDA, Dare MF, Castral TC, Ribeiro LM. Hammock and nesting in preterm infants: randomized controlled trial. Rev Bras Enferm. 2019 Dec;72(suppl 3):96-102. doi: 10.1590/0034-7167-2018-0099. English, Portuguese. PMID 31851240
- [Background] Gerull R, Cignacco E, Stoffel L, Sellam G, Nelle M. Physiological parameters after nonpharmacological analgesia in preterm infants: a randomized trial. Acta Paediatr. 2013 Aug;102(8):e368-73. doi: 10.1111/apa.12288. Epub 2013 May 28. PMID 23651076
- [Background] Huang CM, Tung WS, Kuo LL, Ying-Ju C. Comparison of pain responses of premature infants to the heelstick between containment and swaddling. J Nurs Res. 2004 Mar;12(1):31-40. doi: 10.1097/01.jnr.0000387486.78685.c5. PMID 15136961
- [Background] Schwendener RA, Schott H, Hartmann HR, Supersaxo A, Rubas W, Hengartner H. [Liposomes as carriers of lipophilic cytosine arabinoside and fluorodeoxyuridine derivatives. Their cytostatic effect and possibilities of tumor cell specific therapy]. Onkologie. 1987 Aug;10(4):232-9. doi: 10.1159/000216411. German. PMID 2959889